CLINICAL TRIAL: NCT02869139
Title: Package of Mentholated Measures for the Relief of Thirst in the Anesthesia Recovery Room: Randomized Clinical Trial
Brief Title: Package of Mentholated Measures for the Relief of Thirst in the Anesthesia Recovery Room
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual de Londrina (Other)
Responsible Party: Principal Investigator, Viviane Moreira Serato, Principal Investigator, Master's degree in Nursing, Universidade Estadual de Londrina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GPS Menthol
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Thirst; Mouth Dryness; Irritation Lips
Keywords: Thirst; Ice; Menthol; Perioperative Nursing.; Recovery Room
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Package of mentholated measures (Experimental): Package of mentholated measures (mentholated Ice Popsicle and lip moisturizing) Group.
  Interventions: Other: Mentholated lip moisturizer and ice popsicle
- Package of non-mentholated measures (Active Comparator): Package of non-mentholated measures (mentholated Ice Popsicle and lip moisturizing) Group.
  Interventions: Other: Non-mentholated lip moisturizer and ice popsicle

INTERVENTIONS:
Other: Mentholated lip moisturizer and ice popsicle — Mentholated package of measures
  Arms: Package of mentholated measures
Other: Non-mentholated lip moisturizer and ice popsicle — Non-mentholated package of measures
  Arms: Package of non-mentholated measures

SUMMARY:
Package of mentholated measures for the relief of thirst in the anesthesia recovery room: Randomized clinical trial

DETAILED DESCRIPTION:
Perioperative thirst is intense and has a high incidence. There is evidence that strategies using cold and menthol could be viable alternatives to reduce thirst and the discomforts arising from it. For that reason, this study evaluated the efficacy of a mentholated package of measures (lip moisturizer and ice popsicle) compared to a non-mentholated package of measures in alleviating thirst in the anesthesia recovery room.

ELIGIBILITY:
Inclusion Criteria:

* Possess aged between eighteen and sixty-five years
* To be fasting for more than four hours
* Verbalizing headquarters spontaneously or after questioning, with greater than or equal to three intensity in numerical verbal scale
* Receive opioids or anticholinergic during surgery duration of greater than one hour anesthesia
* Being in anesthetic recovery in anesthesia recovery room
* Have been approved in the evaluation Headquarter Insurance Management Protocol which was applied to both groups
* Accept participate and sign the consent form Clarified

Exclusion Criteria:

* Being allergic to menthol
* Have continuity of injury in the oral mucosa
* Having suspended the anesthetic-surgical procedure after acceptance of participation
* Receive High operating room directly to another healthcare sector than the anesthetic recovery room, and intensive care unit or hospital unit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-04; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Change in intensity of thirst, lip hydration, dryness of the mouth and taste the final oral cavity above the original between the experimental and control groups. | three times: 0 minutes, 30 minutes and 60 minutes after intervention and evaluation
  The evaluation procedures were repeated every 30 minutes for one hour, representing three evaluation moments (M1, M2 and M3).

SECONDARY OUTCOMES:
Change in the extent of satiety point over an hour assessment, presented by experimental and control groups, and the number of interventions required in every moment of assessment and intervention for each group. | three times: 0 minutes, 30 minutes and 60 minutes after intervention and evaluation
  The evaluation procedures were repeated every 30 minutes for one hour, representing three evaluation moments (M1, M2 and M3).

CONTACTS AND LOCATIONS:
Overall Officials: Viviane Serato, Principal Investigator — Universidade Estadual de Londrina
Locations (1):
- Viviane Moreira Serato, Londrina, Paraná, Brazil

IPD SHARING:
Plan to Share IPD: Yes